CLINICAL TRIAL: NCT06451146
Title: Evaluation of the Safety and Efficacy of Orbital Atherectomy (OA) for Calcified Lesions in Patients With Coronary Artery Disease: The Lower Silesian Orbital Atherectomy Registry (LOAR)
Brief Title: Lower Silesian Orbital Atherectomy Registry (LOAR)
Acronym: LOAR
Status: Recruiting | Type: Observational
Sponsor: Regional Cardiology Center, The Copper Health Centre (MCZ), (Other)
Collaborators: Department of Cardiology, Provincial Specialized Hospital in Legnica, 59-200 Legnica, Poland. (Unknown)
Responsible Party: Sponsor
Other Study IDs: CopperHealthCentre4
Record Dates: First submitted 2024-03-03; First posted 2024-06-11 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Safety Issues; Efficacy, Self
Keywords: Percutaneous coronary interventions; Calcified Lesion; Coronary artery diseases; Orbital Atherectomy; Lesion preparation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- OA Intervention: All consecutive patients with moderate/ severely calcified coronary lesions who underwent PCI facilitated by the Orbital Atherectomy The decision to perform orbital atherectomy was left to the operator's dissertation after the detection of a moderate/severely calcified lesion. Angiographic calcification was classified as moderate when it involved between 30% and 50% of the reference lesion diameter, and severe when it occupied over 50% of the reference diameter. When the initial assessment was based on IVUS finding lesion had to reach at least 2 points in the IVUS calcium score. There were no angiographic exclusion criteria regarding lesion anatomy such as the length, tortuosity, severity, or location. All procedural features(use additional lesion preparation technique; stent implantation parameters, periprocedural pharmacological therapy, use of intravascular imaging along with the left ventricular support device) were left to the discretion of the operator.
  Interventions: Procedure: PCI Facilitated with Orbital Atherectomy Device

INTERVENTIONS:
Procedure: PCI Facilitated with Orbital Atherectomy Device — Percutaneous coronary intervention for coronary artery disease supported by the Orbital Atherectomy Device

SUMMARY:
The Lower Silesian Orbital Atherectomy Registry (LOAR), is an observational registry collecting all consecutive cases of percutaneous coronary intervention (PCI) performed with the support of the Orbital Atherectomy Device due to the presence of calcified lesion in coronary arteries. Data will be collected in two cooperating cardiac centers (Department of Cardiology, The Copper Health Center, Lubin, Poland, and Department of Cardiology, Provincial Specialized Hospital in Legnica, Poland).

DETAILED DESCRIPTION:
The study population consisted of all consecutive patients with severely calcified coronary lesions undergoing percutaneous coronary intervention (PCI) with the Orbital Atherectomy Device at two cooperating cardiac centers (Department of Cardiology, The Copper Health Center, Lubin, Poland, and Department of Cardiology, Provincial Specialized Hospital in Legnica, Poland). All study patients had a clinical indication for PCI based on current European Society of Cardiology (ESC) revascularization guidelines, with local heart team support where appropriate.

The decision to perform OA-assisted PCI was left to the discretion of the operator, based on clinical and angiographic features with a concomitant assessment of calcification. Only patients with moderate or severe calcification were enrolled. Calcification severity was defined either by angiographic assessment or by intravascular assessment using intravascular ultrasound (IVUS) and/or optical coherence tomography (OCT). All patients were thoroughly informed about all therapeutic options and PCI-related risks before giving written consent.

ELIGIBILITY:
Inclusion Criteria:

* The presence of moderately to severely calcified lesions.

Exclusion Criteria:

* Lack of patient consent
* Target vessel perforation due to previous unsuccessful lesion preparation
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of all consecutive patients from the two cooperating cardiology departments in the Lower Silesia region with a clinical indication for PCI and the presence of severely calcified lesions who underwent percutaneous coronary intervention facilitated by an orbital atherectomy device. The decision to perform orbital atherectomy was left to the operator after detection of a moderate/severely calcified lesion.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
The rate of patients who achieved The Clinical Success | Evaluation at discharge (assessed up to day 10)
  Clinical success was defined as effective stent deployment without significant stent under expansion and the presence of Thrombolysis in Myocardial Infarction (TIMI) 3 flow at the end of the procedure.
Incidence of Treatment-Emergent Adverse Events | Evaluation at discharge (assessed up to day 10)
  The safety outcomes were defined as procedural complications(coronary perforation, slow- or no-reflow, new coronary thrombus, ventricular arrhythmias, vessel closure, and device failure).

SECONDARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE) | Final assessment - 5 years after the initial hospitalization; followed by evaluation every 6 months from the end of the hospitalization until the final assessment (5 years)
  MACCE was defined as acute coronary syndrome, cerebrovascular events, major bleeding, need for repeated revascularization, or death.

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Department of Cardiology, Provincial Specialized Hospital in Legnica, Legnica, Lower Silesian Voivodeship
  - Department of Cardiology, The Copper Health Centre (MCZ), Lubin, Lower Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rola P, Kulczycki JJ, Barycki M, Wlodarczak S, Furtan L, Kedzierska M, Giniewicz K, Doroszko A, Lesiak M, Wlodarczak A. Comparison of Orbital Atherectomy and Rotational Atherectomy in Calcified Left Main Disease: Short-Term Outcomes. J Clin Med. 2023 Jun 13;12(12):4025. doi: 10.3390/jcm12124025. PMID 37373718
- [Result] Rola P, Furtan L, Wlodarczak S, Jastrzebski A, Barycki M, Kedzierska M, Szudrowicz M, Kulczycki JJ, Doroszko A, Lesiak M, Wlodarczak A. Orbital atherectomy for treatment of calcified coronary artery lesions. First experiences in Poland: Short-term outcomes of the Lower-Silesia Orbital Atherectomy Registry (LOAR). Kardiol Pol. 2023;81(2):174-176. doi: 10.33963/KP.a2023.0003. Epub 2023 Jan 3. No abstract available. PMID 36594531
- [Result] Rola P, Wlodarczak S, Barycki M, Furtan L, Jastrzebski A, Kedzierska M, Doroszko A, Lesiak M, Wlodarczak A. Safety and Efficacy of Orbital Atherectomy in the All-Comer Population: Mid-Term Results of the Lower Silesian Orbital Atherectomy Registry (LOAR). J Clin Med. 2023 Sep 8;12(18):5842. doi: 10.3390/jcm12185842. PMID 37762782
- [Result] Wlodarczak S, Rola P, Furtan L, Barycki M, Szudrowicz M, Kulczycki JJ, Doroszko A, Lesiak M, Wlodarczak A. Orbital-Tripsy - orbital atherectomy facilitated by Shockwave Intravascular Lithotripsy: Novel bailout strategy in percutaneous coronary intervention in heavily calcified coronary lesions. Kardiol Pol. 2023;81(3):296-297. doi: 10.33963/KP.a2023.0005. Epub 2022 Dec 27. No abstract available. PMID 36573605